CLINICAL TRIAL: NCT00505817
Title: GnRH Agonist and Antagonists in an Oocyte Donation Program
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None
Other Study IDs: VLC-MM-0706-307-19
Record Dates: First submitted 2007-07-23; First posted 2007-07-25 (Estimated); Last update posted 2009-01-12 (Estimated); Status verified 2009-01

CONDITIONS: Effect of Two Protocols of Ovarian Stimulation on Oocyte Quality
MeSH Terms: interventions — cetrorelix; Leuprolide

INTERVENTIONS:
Drug: Cetrorelix and Leuprolide

SUMMARY:
The primary purpose of this study is to evaluate the effect of the two different protocols (long protocol vs antagonist protocol) on oocyte / embryo quality.

DETAILED DESCRIPTION:
The cycles with antagonists of the GnRHa present a series of advantages with respect the GnRHa in an oocyte donation program: treatment cycles are simpler and shorter, a lower amount of dose of gonadotrophins is needed for stimulation, and most important, a decreased rate of ovarian hyperstimulation syndrome is observed. Nevertheless, several clinical trials relate their use to a greater rate of abortion and worse oocyte/ embryo quality. In order to discriminate the endometrial factor from the quality of oocyte cohort, the best strategy is the oocyte donation model. In the present study, for the first time, the effect of different protocols (long versus antagonist protocol) will be studied in the same donor, acting as its own control, undergoing COH. We will compare the COH´s parameters and IVF outcome obtained in the same donor submitted to, firstly, GnRH antagonist protocol (Cetrorelix- n= 45) versus another consecutive cycle with long protocol (Ac. Leuprolide- n= 45).

ELIGIBILITY:
Inclusion Criteria:

* oocyte donors with age range: 18 - 34; BMI: 18 - 29 kg/m2;

Exclusion Criteria:

* PCO

Ages: 18 Years to 34 Years | Sex: Female
Age Groups: Adult

CONTACTS AND LOCATIONS:
Overall Officials: Marco Melo, MDPhD, Principal Investigator — Instituto Valenciano de Infertilidad
Locations (1):
- Instituto Valenciano de Infertilidad Spain, Valencia, Valencia, Spain